CLINICAL TRIAL: NCT04332094
Title: Pilot, Randomized, Multicenter, Open-label Clinical Trial of the Use of Tocilizumab for Treatment of SARS-CoV-2 Infection (COVID-19)
Brief Title: Clinical Trial of the Use of Tocilizumab for Treatment of SARS-CoV-2 Infection (COVID-19)
Acronym: TOCOVID
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Collaborators: Instituto de Salud Carlos III (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIBSP-COV-2020-23
Record Dates: First submitted 2020-03-31; First posted 2020-04-02 (Actual); Last update posted 2021-05-06 (Actual); Status verified 2021-05

CONDITIONS: COVID-19
Keywords: Tocilizumab
MeSH Terms: conditions — COVID-19 | interventions — tocilizumab; Hydroxychloroquine; Azithromycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Early administration of tocilizumab associated with hydroxychloroquine and azithromycin.
  Interventions: Drug: Tocilizumab; Drug: Hydroxychloroquine; Drug: Azithromycin
- Control (Active Comparator): Treatment of SARS-COV-2 (COVID-19) infection with hydroxychloroquine and azithromycin.
  Interventions: Drug: Hydroxychloroquine; Drug: Azithromycin

INTERVENTIONS:
Drug: Tocilizumab — 162 mg sc x 2 doses + tocilizumab 162mg sc x 2 doses at 12 hours (day 1)
  Arms: Intervention
Drug: Hydroxychloroquine — 400 mg / 12h v.o. day 1 followed by 200 mg / 12h v.o. for 6 days (7 days in total)
Drug: Azithromycin — 500 mg / day v.o. for 3 days

SUMMARY:
COVID-19 is a respiratory disease caused by the new coronavirus (SARS-CoV-2) and causes considerable morbidity and mortality.

Currently, there is no vaccine or therapeutic agent to prevent and treat a SARS-CoV-2 infection. This clinical trial is designed to evaluate the use of Tocilizumab in combination with hydroxychloroquine and azithromycin for the treatment of hospitalized adult patients with COVID-19.

ELIGIBILITY:
Inclusion Criteria:

* Subject (or authorized legal representative) who can provide written informed consent before beginning any study procedure.
* Understand and agree to abide by the study procedures.
* Adult #18 years of age at the time of inclusion in the study.
* Confirmation of SARS-CoV-2 infection by a microbiological test performed before randomization, no longer than 72 hours.
* Severity 3-4 according to the WHO 7-point ordinal scale.

Exclusion Criteria:

* ALT / AST> 5 times the normal limit
* Stage 4 chronic kidney disease (GFR <30) or requiring dialysis.
* Presence of comorbidities that imply a poor prognosis (according to clinical judgment).
* Advanced dementia.
* Pregnancy or breastfeeding.
* Anticipation of transfer to another center in the 12 hours at the beginning of the study.
* Allergy to study medication.
* Serious or active bacterial infections or documented sepsis by pathogens other than SARS-CoV-2.
* Streptococcus pneumoniae antigenuria positive before study start.
* Neutropenia <500 / mm3.
* Thrombocytopenia <100,000 / mm3.
* History of diverticulosis.
* Ongoing skin infection (eg, pyodermitis).
* Transplanted patient under immunosuppressive treatment.
* Previous evidence of latent untreated tuberculosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 276 (Estimated)
Dates: Start 2020-04-02 (Actual); Primary Completion 2021-06 (Estimated); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
In-hospital mortality | Through hospitalization, an average of 2 weeks
Need for mechanical ventilation in the Intensive Care Unit | Through hospitalization, an average of 2 weeks

CONTACTS AND LOCATIONS:
Locations (7):
- Spain (7):
  - Hospital Universitario Central de Asturias, Oviedo, Principality of Asturias
  - Hospital General Universitario de Alicante, Alicante, Valencia
  - Hospital General Universitario de Elche, Elche, Valencia
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital del Mar, Barcelona
  - Hospital Sant Joan Despí, Barcelona
  - Hospital Clinico San Carlos, Madrid